CLINICAL TRIAL: NCT01813253
Title: A Randomized, Open-label, Japan-Korea-Taiwan Collaborative Phase 3 Study to Compare the Efficacy of Nimotuzumab and Irinotecan Combination Therapy Versus Irinotecan Monotherapy as Second Line Treatment in Subjects With Advanced or Recurrent Gastric and Gastroesophageal Junction Cancer
Brief Title: Phase 3 Study of Nimotuzumab and Irinotecan as Second Line With Advanced or Recurrect Gastric and Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DE766-A-J302
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: epidermal growth factor receptor; second line
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irinotecan and nimotuzumab (Experimental): Adminitration of irinotecan 150 mg/m2 IV once every 2 weeks and nimotuzumab 400 mg IV once weekly
  Interventions: Drug: Irinotecan; Drug: Nimotuzumab
- Irinotecan (Active Comparator): Administration of irinotecan 150 mg/m2 IV once every 2 weeks
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — 150 mg/m2 IV once every 2 weeks until progression or unacceptable toxicity develops
  Other Names: Boryung irinotecan
Drug: Nimotuzumab — 400mg IV once weekly until progression or unacceptable toxicity develops
  Other Names: DE-766
  Arms: Irinotecan and nimotuzumab

SUMMARY:
This study will evaluate overall survival of nimotuzumab in combination with irinotecan compared to irinotecan alone in subjects with EGFR overexpressed advanced gastric or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
This randomized, open-label, Japan, Korea and Taiwan collaborative, phase 3 study will evaluate overall survival of nimotuzumab in combination with irinotecan compared to irinotecan alone in subjects with EGFR overexpressed advanced gastric or gastroesophageal junction cancer. Approximately 400 subjects will be randomized in a 1:1 ratio to receive irinotecan (control group) or nimotuzumab and irinotecan (combination group). Nimotuzumab and/or irinotecan should be continued until disease progression or intolerable toxicity. Nimotuzumab is administered at 400 mg once weekly as an intravenous infusion and irinotecan is administered at 150 mg/m2 once every 2 weeks as an intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or recurrent subjects with gastric or gastroesophageal junction adenocarcinoma.
2. Subjects who experienced disease progression during first line or within 6 months after the last dose of first line therapy. The first line regimen must have contained a 5-fluorouracil based agent and platinum agent.
3. Subjects with EGFR overexpression (2+ or 3+ in IHC)

Exclusion Criteria:

1. Subjects who have received irinotecan
2. Subjects who have received EGFR-directed therapy
3. Other active malignancy within the last 5 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Around 4.5 years after first subject randomization
  Overall survival is defined as the time from the date of randomization to the date of the death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival | Around 4.5 years after first subject randomization
  Progression Free Survival is defined as the time from the date of randomization to the date of progression or death from any cause, whichever comes first.
Overall Response Rate | Around 4.5 years after first subject randomization
  Overall Response Rate is defined as the proportion of subjects with CR or PR in the best overall response.
Disease Control Rate | Around 4.5 years after first subject randomization
  Disease Control Rate is defined as the proportion of subjects with CR, PR or SD in the best overall response.
Incidence of adverse events | Around 4.5 years after first subject randomization
  Incidence of adverse events using latest CTCAE version 4 including minor version

CONTACTS AND LOCATIONS:
Locations (36):
- Japan (22):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Aichi
  - Akita
  - Aomori
  - Chiba
  - Ehime
  - Fukuoka
  - Hiroshima
  - Hokkaido
  - Hyōgo
  - Ishikawa
  - Kanagawa
  - Kumamoto
  - Kyoto
  - Nagano
  - Niigata
  - Osaka
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokyo
  - Toyama
- South Korea (9):
  - Busan
  - Daegu
  - Hwansun Junnam hospital, Gwangju
  - Gyeonggi-do
  - Incheon
  - Jeonju
  - Seongnam
  - Seoul
  - Yangsan
- Taiwan (5):
  - Changhua
  - Tainan
  - Taipei
  - Taoyuan District
  - Thaichung